CLINICAL TRIAL: NCT06679556
Title: A Phase 1 Randomized, Double Blind, Crossover Pharmacokinetic Study of Minoxidil Sublingual Tablets in Adult Male and Female Healthy Volunteers.
Brief Title: Phase 1 Pharmacokinetic Study of Minoxidil SL Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samson Clinical Operations Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SAM-001
Record Dates: First submitted 2024-10-21; First posted 2024-11-07 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pharmacokinetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strength A Sublingual Minoxidil (Experimental)
  Interventions: Drug: Strength A Sublingual Minoxidil
- Strength B Sublingual Minoxidil (Experimental)
  Interventions: Drug: Strength B Sublingual Minoxidil

INTERVENTIONS:
Drug: Strength A Sublingual Minoxidil — One single dose of Strength A sublingual minoxidil
  Arms: Strength A Sublingual Minoxidil
Drug: Strength B Sublingual Minoxidil — One single dose of Strength B sublingual minoxidil
  Arms: Strength B Sublingual Minoxidil

SUMMARY:
This is a phase 1 randomized, double blind, crossover study examining the pharmacokinetic profile of two different doses of minoxidil sublingual tablets in healthy adult volunteers.

The main objective is to determine the pharmacokinetics of minoxidil following sublingual administration of a single dose in adult male and female healthy volunteers. The secondary objective is to evaluate the safety of minoxidil following sublingual administration of a single dose in adult male and female healthy volunteers.

A total of 12 participants (6 male and 6 female) will be recruited for study participation.

The duration of study participation is up to 43 days including screening and safety follow up. A single dose of study medication (strength A or strength B) will be administered on Day 1 to all study participants and PK samples will be taken periodically over a 12-hr period. After at least 7-day washout period the other dose of study medication (strength B or strength A, respectively) will be administered to all participants and PK samples will be taken periodically over a 12-hr period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 65 years of age (inclusive) at screening.
* In good general health in the opinion of the Investigator based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring (ECG). A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if, in the opinion of the Investigator, the finding is (a) unlikely to introduce additional risk to the subject, (b) will not interfere with study procedures or confound study results, and (c) is not listed in the Exclusion Criteria.
* Body mass index (BMI) is between 18.5 - 30.0 kg/m2 with a body weight of at least 50 kg.
* Have systolic blood pressure within normal limits (90-140 mm Hg).
* Have adequate venous access on their left or right arm to allow collection of multiple blood samples.
* Women of Childbearing Potential (WOCBP) must agree to use a highly effective method of contraception from enrolment to the safety follow-up visit.
* Women of non-childbearing potential must be post-menopausal or permanently sterilised at least 6 months prior to screening.
* All WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test before dosing on each dosing day.
* Willing and able to attend all study visits and comply with treatment plan and required study procedures.
* Able to comprehend and willing to sign and date a written informed consent form.

Exclusion Criteria:

* History of hypersensitivity or allergies to any ingredients contained in the study medication.
* A positive urine drugs of abuse screen at Screening or alcohol breath test on dosing days, unless for a legitimate medical reason as determined by the Investigator.
* A positive Hepatitis B surface antigen, Hepatitis C antibody result, or human immunodeficiency virus (HIV) result at screening.
* Current participation in any other investigational drug or medical device trial, which includes administration of an investigational study medication or medical device, or within 3 months or 5 half-lives of the investigational product, whichever is longer, prior to receiving first dose.
* Unwilling to comply with all study procedures and assessments.
* Participants with specific underlying conditions (e.g. cardiovascular disease, cardiac arrhythmia, hepatic comorbidity, renal comorbidity, phaeochromocytoma), clinically significant findings from medical history, clinical laboratory tests, ECG, or vital signs that, in the opinion of the Investigator, could interfere with the objectives of the study or put the participant at risk.
* Use of anti-hypertensive medication or any other medications that, in the opinion of the Investigator, could interfere with the objectives of the study or put the participant at risk, within 14 days or 5 half-lives (whichever is longer) before the start of the study treatment.
* A history of alcoholism, substance or drug abuse-related disorders in the past year as deemed significant by the Investigator.
* Pregnant, planning a pregnancy, or nursing a child.
* Major surgery within 4 weeks prior to the screening evaluation, or planned surgery prior to completion of all study procedures.
* Donation of blood or blood products of 470 mL or greater within 12 weeks prior to dosing in Period 1.
* Dietary requirements that prevent consumption of the standardised study meals.
* Poor complier or unlikely to attend specified study days.
* Study site or Sponsor employee, or immediate family member of a study site or Sponsor employee.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time profile (AUClast, AUCinf) of sublingual minoxidil | At Day 1 and Day 8
  The primary endpoints will be the area under the concentration-time curve from time zero to the last measurable concentration (AUClast), the area under the concentration-time curve from time zero to infinity (AUCinf), maximum concentration (Cmax), time to maximum concentration (Tmax), half-life (T1/2), and the terminal rate constant (λz).
  AUClast measures the total minoxidil exposure in the body up to the last measurable time point, while AUCinf estimates total minoxidil exposure from the time it's taken until it completely leaves the body.
Maximum observed concentration (Cmax) of sublingual minoxidil | At Day 1 and Day 8
  The primary endpoints will be the area under the concentration-time curve from time zero to the last measurable concentration (AUClast), the area under the concentration-time curve from time zero to infinity (AUCinf), maximum concentration (Cmax), time to maximum concentration (Tmax), half-life (T1/2), and the terminal rate constant (λz).
  Cmax is the highest concentration of minoxidil in the blood after it's taken.
Time of maximum observed concentration (Tmax) of sublingual minoxidil | At Day 1 and Day 8
  The primary endpoints will be the area under the concentration-time curve from time zero to the last measurable concentration (AUClast), the area under the concentration-time curve from time zero to infinity (AUCinf), maximum concentration (Cmax), time to maximum concentration (Tmax), half-life (T1/2), and the terminal rate constant (λz).
  Tmax measures the time it takes for minoxidil to reach its highest concentration in the blood after it's taken.
Terminal rate constant (λz) of sublingual minoxidil | At Day 1 and Day 8
  The primary endpoints will be the area under the concentration-time curve from time zero to the last measurable concentration (AUClast), the area under the concentration-time curve from time zero to infinity (AUCinf), maximum concentration (Cmax), time to maximum concentration (Tmax), half-life (T1/2), and the terminal rate constant (λz).
  The terminal rate constant measures the speed at which the concentration of minoxidil decreases in the blood during the last stage of elimination.
Terminal half-life (T½) of sublingual minoxidil | At Day 1 and Day 8
  The primary endpoints will be the area under the concentration-time curve from time zero to the last measurable concentration (AUClast), the area under the concentration-time curve from time zero to infinity (AUCinf), maximum concentration (Cmax), time to maximum concentration (Tmax), half-life (T1/2), and the terminal rate constant (λz).
  The terminal half-life measures the time it takes for the concentration of minoxidil in the blood to decrease by half during the last stage of elimination.

SECONDARY OUTCOMES:
Type of adverse events | At Day 1, Day 8, and Day 15
  The safety profile of sublingual minoxidil will be evaluated by analyzing the type, incidence, relationship to study drug and severity of adverse events for each dose of sublingual minoxidil. It will also be evaluated through the change from baseline in clinical safety monitoring parameters, including clinical laboratory tests, vital signs, and ECG.
Incidence of Adverse Events | At Day 1, Day 8, and Day 15
  The safety profile of sublingual minoxidil will be evaluated by analyzing the type, incidence, relationship to study drug and severity of adverse events for each dose of sublingual minoxidil. It will also be evaluated through the change from baseline in clinical safety monitoring parameters, including clinical laboratory tests, vital signs, and ECG.
Relationship of adverse events to study drug | At Day 1, Day 8, and Day 15
  The safety profile of sublingual minoxidil will be evaluated by analyzing the type, incidence, relationship to study drug and severity of adverse events for each dose of sublingual minoxidil. It will also be evaluated through the change from baseline in clinical safety monitoring parameters, including clinical laboratory tests, vital signs, and ECG.
Severity of adverse events | At Day 1, Day 8, and Day 15
  The safety profile of sublingual minoxidil will be evaluated by analyzing the type, incidence, relationship to study drug and severity of adverse events for each dose of sublingual minoxidil. It will also be evaluated through the change from baseline in clinical safety monitoring parameters, including clinical laboratory tests, vital signs, and ECG.
Change from baseline in clinical safety monitoring parameters | At Day 1, Day 8, and Day 15
  The safety profile of sublingual minoxidil will be evaluated by analyzing the type, incidence, relationship to study drug and severity of adverse events for each dose of sublingual minoxidil. It will also be evaluated through the change from baseline in clinical safety monitoring parameters, including clinical laboratory tests, vital signs, and ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Rodney Sinclair Pty Ltd, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No